CLINICAL TRIAL: NCT06056154
Title: Safety and Efficacy of the Hydrophobic Intraocular Lens Asqelio Monofocal With Biaspheric Design
Status: Enrolling by invitation | Type: Observational
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQM012023
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cataract; Pseudophakia
MeSH Terms: conditions — Cataract; Pseudophakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing routine clinical practice with ASQELIOTM monofocal LIO model QLIO130C.: Data will be extracted retrospectively from their medical records and prospectively in a single follow-up visit. All procedures performed are according to standard clinical practice.
  Interventions: Device: LIO ASQELIO TM monofocal QLIO130C

INTERVENTIONS:
Device: LIO ASQELIO TM monofocal QLIO130C — Intraocular lens (IOL) implant. All patients will have been treated as per standard clinical practice.

SUMMARY:
The goal of this observational study is to learn about the Asqelio monofocal intraocular lens (IOL) model QLIO130C in patients undergoing cataract surgery. The aim of the study is to evaluate the lens implementation safety and efficacy after at least 24 months.

DETAILED DESCRIPTION:
This is a retro-prospective, post-marketing observational study of a CE-marked medical device. The efficacy and safety of the Asqelio monofocal intraocular lens (IOL) model QLIO130C from AST Products, Inc, Billerica, USA, will be studied in patients implanted according to standard clinical practice. Twelve-month follow-up data will be collected from the medical records of the patients included in the study, and after 24 months they will be scheduled for a review.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 22 years of age or older undergoing cataract surgery in at least 1 eye and implanted with ASQELIO monofocal model QLIO130C.
* Subjects for whom postoperative emmetropia (±0.5 D spherical equivalent) was planned.

Exclusion Criteria:

* Any pathology that reduces the potential Visual Acuity (VA) with its best correction beyond 0.30 logMAR.
* Previous corneal surgery.
* Rubella or surgery due to traumatic cataract.
* Ocular trauma or refractive surgery.
* Any other ocular or systemic condition that, in the opinion of the investigator, should exclude the subject from the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects undergoing cataract surgery, implanted with ASQELIO monofocal model QLIO130C, and with a follow-up of more than 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Posterior capsular opacity | 24 months after IOL implantation
  Incidence of PCO
Intensity of Posterior capsular opacity | 24 months after IOL implantation
  Intensity of PCO determined using LOCSIII Classification
Visual acuity | At least 24 months after IOL implantation
  Best corrected distance visual acuity in LogMAR units using the ETDRS chart

SECONDARY OUTCOMES:
Refraction | At least 24 months after IOL implantation
  Residual refractive error in diopters determined objectively
Incidence of Glistening | At least 24 months after IOL implantation
  Incidence of IOL glistening
Intensity of Glistening | 24 months after IOL implantation
  Intensity of IOL glistening. It will be evaluated by examining the center of the IOL optical zone with the pupil dilated using a slit lamp. The intensity of glistening will be graded as the number of glistening in the central region according to the following scale: 0 = absent, 1 = traceable (countable vacuoles), 2=moderate (low density of countless vacuoles), and 3=severe (high density of countless vacuoles).

CONTACTS AND LOCATIONS:
Locations (1):
- Oftalmología Vistahermosa SL, Alicante, Spain